CLINICAL TRIAL: NCT01719588
Title: A Post-Marketing Surveillance (PMS) Study on the Safety and Effectiveness of Prolonged Release Tapentadol Hydrochloride Among Adult Filipino Patients With Moderate To Severe Chronic Non-Cancer Pain
Brief Title: A Safety and Effectiveness Study of Prolonged Release Tapentadol Hydrochloride Among Filipino Patients With Moderate to Severe Chronic Non-Cancer Pain
Status: Withdrawn | Type: Observational
Why Stopped: The company decided to cancel this study in conformity with PH FDA Circular 2013-004
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100918; R331333PAI4007 (Other: Janssen Pharmaceutica); TPD-C-12-PH-001-V02 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Moderate to Severe Chronic Non-cancer Pain
Keywords: Moderate to severe chronic non-cancer pain; Prolonged release tapentadol hydrochloride; Tapentadol PR; Extended release tapentadol hydrochloride; Nucynta PR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prolonged release tapentadol: Patients will be taking prolonged release tapentadol hydrochloride as per the product insert approved in Philippines.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Prolonged release tapentadol hydrochloride will be administered as per the recommended doses approved in Philippines. The recommended oral starting dose is 50 mg, 100 mg, 150 mg, 200 mg, or 250 mg every 12 hours, with or without food depending on the initial pain intensity and thereafter, the dose will be adjusted to maintain adequate analgesia with acceptable tolerability. The dosing regimen will be individualized according to the severity of pain being treated, the previous treatment experience, and the ability to monitor patients.
  Other Names: Nucynta PR

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of prolonged release tapentadol hydrochloride for the relief of moderate to severe chronic non-cancer pain among Filipino patients.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-center (study conducted at multiple sites), observational study (study in which the investigators/ physicians observe the patients and measure their outcomes). The study will enroll approximately 100 patients who will be taking prolonged release tapentadol hydrochloride with a dosing regimen stipulated in the product insert. As this is an observational study, assessment of patient will be based on the accepted clinical practice in the Philippines. Patients will be monitored at baseline (Day 1) and throughout the 84-day treatment period of prolonged release tapentadol hydrochloride (every 7 days for the first two weeks, and thereafter every 28 days for the next three months) for effectiveness with the help of short form Brief Pain Inventory (BPI) questionnaire. Safety evaluations will include assessment of adverse events, clinical laboratory tests, and co-morbid conditions. The total study will be conducted for 3 years and the duration of treatment will be for 84 days.

ELIGIBILITY:
Inclusion Criteria:

* Filipino patients with moderate to severe non-cancer pain with an onset of 12 weeks or less from the baseline visit and pain requires Schedule 2 opioid treatment as per assessment of the prescribing physician
* Patients who able to independently communicate pain characteristics, understand and complete self administered questionnaires
* Medically stable on the basis of routine physical examination, medical history, and vital signs at the time of baseline visit

Exclusion Criteria:

* Refuse to protocol-defined use of effective contraception
* Pregnant and lactating women
* Patients with severe renal and hepatic impairment, significant respiratory depression, acute or severe bronchial asthma or hypercapnia, and having or suspected paralytic ileus
* Patients with acute intoxication with alcohol, hypnotics, centrally acting analgesics, or psychotropic drugs or receiving other mu-opioid receptor agonist analgesics, general anesthetics, phenothiazines, other tranquilizers, and sedatives
* Patients who are receiving Monoamine oxidase (MAO) inhibitors or who have taken them within the last 14 days
* Patients with documented history of increased intracranial pressure, impaired consciousness, coma and seizure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino patients with moderate to severe chronic non-cancer pain and who are on the approved product label of prolonged release tapentadol hydrochloride
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients with incidence of adverse events and adverse drug reactions | From the date of first exposure of patient to the study medication until 30 days after the last dose of the study medication and at anytime the investigator deems it as necessary, as assessed for 3 years

SECONDARY OUTCOMES:
The short form Brief Pain Inventory (BPI) questionnaire scores | Baseline (Day 1), Day 7, Day 14 and Day 28, Day 56, and Day 84
  The short form BPI allows patients to rate the severity of their pain on a scale of 0 (no pain) to 10 (pain as bad as you can imagine) and the degree to which their pain interferes with common dimensions of feeling and function (general activity, walking, work, mood, enjoyment of life, relations with others, and sleep) on a scale of 0 (no interference) to 10 (interferes completely).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica